CLINICAL TRIAL: NCT02356341
Title: NovaTears® Observational Study NT-002
Brief Title: NovaTears® Eye Drops Observational Study NT-002
Status: Completed | Type: Observational
Sponsor: Novaliq GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: NT-002
Record Dates: First submitted 2015-01-21; First posted 2015-02-05 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NovaTears®
  Interventions: Device: NovaTears® Eye Drops

INTERVENTIONS:
Device: NovaTears® Eye Drops — Topical eye drops for lubrication of the ocular surface

SUMMARY:
This observational study is intended to collect outcome data from a cohort of 90 patients suffering from symptoms of dry eye disease due to meibomian gland dysfunction who are treated with the medical device NovaTears® eye drops for a duration of 6 to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* According to NovaTears® instruction for use
* ≥ 18 years
* Patients with dry eye disease due to meibomian gland dysfunction applying eye lid hygiene for at least 14 days
* Ability and willingness to provide written Informed Consent
* Ability and willingness to participate in all examinations
* Willingness and ability to return for follow up visit

Exclusion Criteria:

* Patients with hypersensitivity to any of the components of NovaTears®
* Patients with contact lenses, pregnancies, or who are breast feeding
* Patients with dry eye disease not caused by meibomian gland dysfunction
* Patients taking lipid containing eye drops or requiring topical pharmacological treatment of dry eye disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with dry eye disease due to meibomian gland dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Subjective symptom severity | 6 to 8 weeks
  Change in subjective symptom severity score compared to Baseline

SECONDARY OUTCOMES:
Tear-Film Break-up Time | 6 to 8 weeks
  Change in Tear Film Break-up Time (measured in seconds) compared to Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Novaliq GmbH, Study Director — Novaliq GmbH
Locations (8):
- Germany (8):
  - Prof. Dr. Norbert Schrage, Cologne
  - University Eye Hospital of the HHU Duesseldorf, Düsseldorf
  - University Eye Hospital of the FAU Erlangen-Nuremberg, Erlangen
  - University Eye Hospital Heidelberg, Heidelberg
  - Dr. Thomas Kaercher, Heidelberg
  - JenVis Research Institute, Jena
  - Staedtisches Klinikum Karlsruhe, Karlsruhe
  - University Eye Hospital, LMU Munich, Munich

REFERENCES:
- [Derived] Steven P, Augustin AJ, Geerling G, Kaercher T, Kretz F, Kunert K, Menzel-Severing J, Schrage N, Schrems W, Krosser S, Beckert M, Messmer EM. Semifluorinated Alkane Eye Drops for Treatment of Dry Eye Disease Due to Meibomian Gland Disease. J Ocul Pharmacol Ther. 2017 Nov;33(9):678-685. doi: 10.1089/jop.2017.0042. Epub 2017 Sep 18. PMID 28922088